CLINICAL TRIAL: NCT01355731
Title: Evaluating Therapeutic Boundaries Among Bedside Nurses At A Pediatric Hematology/Oncology Research Hospital
Acronym: EBABN
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XMP10-163 ETBABN
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Last update posted 2011-09-15 (Estimated); Status verified 2011-09

CONDITIONS: Therapeutic Boundaries; Nurse-Patient Relations
Keywords: Registered Nurse; Behaviors; Attitudes
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Registered Nurse: This is quality improvement study that is descriptive and is utilizing a convenience sample of direct care registered nurses employed full-time for at least one year at St. Jude Children's Research Hospital.Participants will take a onetime researcher generated therapeutic boundaries questionnaire which will describe behaviors and attitudes regarding therapeutic boundaries.

SUMMARY:
Professional therapeutic boundaries are defined as the limits that protect the space between a professional's power and patient's vulnerability. It is important to develop therapeutic alliances while maintaining boundaries, thus ensuring nurses develop safe connections with patients and their families based on therapeutic needs. Due to the professional nature of nursing, boundary violations are common. For example, closeness and familiarity develops between the healthcare provider, patient, and caregiver that encompass the physical, emotional, and spiritual realms. This provides an opportunity for intense bonds with patients and families. Furthermore in oncology healthcare, providers deliver compassionate care and empathize with patients and families while sharing in the patient's illness journey. As a result of these bonds and relationships the nurse may over disclose personal information, provide excessive patient attention, meeting their own personal needs instead of the patient and family. In addition, continuity of care contributes to boundary crossings because there is frequent repeated contact with the same patients and families which allows blurring of boundary lines. When staff spend weeks, months, or even years with the same patient the opportunity to connect and talk about personal life details exist. At the national level, the National Council of State Boards of Nursing (NCSBN) has created materials for educating nurses in maintenance of therapeutic boundaries. Adherence to therapeutic boundaries has now become an education objective, with the development of educational interventions within many health care settings. Likewise, St. Jude nurses are at an increased risk of crossing therapeutic boundaries due to long term care relationships and vulnerable family members. However, nursing administration has not formally assessed the attributes or behaviors of the nursing staff. This proposal will describe the attributes and behaviors of the St. Jude staff nurse towards nurse-patient/family boundaries, providing knowledge to nursing leadership that will facilitate therapeutic boundaries focus groups with direct care nurses.

DETAILED DESCRIPTION:
Participants will take a onetime researcher generated therapeutic boundaries questionnaire which will describe behaviors and attitudes regarding therapeutic boundaries.

The main objective of the study is to :

To describe behaviors and attitudes towards nurse-patient/family boundaries of direct patient care Registered Nurses (RNs) at St. Jude Children's Research Hospital

ELIGIBILITY:
Inclusion Criteria:

* Registered Nurse (RN)
* Employed at St. Jude Children's Research Hospital at least one year
* Employed full-time (at least 90% full-time equivalent - works at least 72 hours every two weeks).
* provides direct patient care

Exclusion Criteria:

Declines survey participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is quality improvement study that is descriptive and is utilizing a convenience sample of direct care registered nurses employed full-time for at least one year at St. Jude Children's Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2011-05; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Behaviors and attitudes of nurse-patient/family boundaries among registered nurses (RNs) at St. Jude Children's Research Hospital that provide direct patient care. | 6 months
  Each question will be analyzed and interpreted individually. More importantly, for each question, the percentage of nurses reporting "sometimes" or "often" will be reported because the questions where nurses more likely to score high are good references for planning the future nursing education series.

CONTACTS AND LOCATIONS:
Overall Officials: La-Kenya Kellum, DNP, RN, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org